CLINICAL TRIAL: NCT00107614
Title: UARK 2002-10, A Phase II Study of DT PACE Induction, Followed by Tandem Autologous Transplant and Maintenance Therapy for Patients With Advanced and/or Symptomatic Waldenstrom's Macroglobulinemia
Brief Title: DT PACE, Tandem Autologous Transplant, Maintenance Therapy for Waldenstrom's Macroglobulinemia Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to poor accrual.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UARK 2002-10
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Results first posted 2011-07-15 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: Waldenstrom
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DT PACE/auto transplant/maint therapy (Experimental)
  Interventions: Drug: DT PACE + Rituxan

INTERVENTIONS:
Drug: DT PACE + Rituxan — INDUCTION PHASE DT PACE + Rituxan DT PACE + Rituxan + PBSC Collection Response Assessment TRANSPLANT PHASE Transplant 1 (MEL 200 (patients with < 50% response to induction) OR MEL-DT PACE (Patients with > 50% response to Induction) Transplant 2 (identical to the first, except patients with progressive or proliferative disease, will receive BEAM) MAINTENANCE PHASE Rituxan every 3 months x 1 year

SUMMARY:
The purpose of this study is to find out what the response is and the side effects are with chemotherapy using a combination of drugs called D.T. PACE (Dexamethasone, Thalidomide, cis-Platinum, Adriamycin, Cyclophosphamide, and Etoposide) + Rituxan, followed by two autologous transplants.

DETAILED DESCRIPTION:
Approximately 25 patients, male or female, age 18 and older, regardless of race or ethnicity, will participate in this study at UAMS (University of Arkansas for Medical Sciences) only.

Participants will receive two courses of chemotherapy with a regimen called DT PACE + Rituxan. This regimen consists of 6 drugs: Dexamethasone, Thalidomide, cis-Platinum, Adriamycin, Cyclophosphamide, and Etoposide.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathological diagnosis of Waldenstrom's Macroglobulinemia, with advanced and/or symptomatic disease requiring therapy. At least one of the following must be true: *Presence of cytopenias, defined as Hemoglobin < 11 gm%, or WBC < 2000/µl, or platelets < 100,000 µl; *Presence of extensive (>3 cm) or symptomatic lymphadenopathy or hepatosplenomegaly; *Presence of B symptoms (night sweats, fever, weight loss of >10% of the baseline); *Presence of severe neuropathy, not otherwise explained; *Progressive disease (increase in "M" by > 50% while observed, and decrease in hemoglobin by >2 gm%,and/or decrease in platelets by >50,000/µl, and/or increase in lymphadenopathy); *Serum albumin <2.5 gm%; *Persistently elevated β-2M >3.0 in the absence of renal impairment or active infection.
* Hyperviscosity will be treated (in addition to plasmapheresis) only in the presence of any of the above
* All necessary baseline studies for determining eligibility must be obtained within 35 days prior to registration.
* Patients must have a performance status of 0-2 based on SWOG criteria. Patients with a poor performance status (3-4), based solely on bone pain, will be eligible.
* Patients must not have significant co-morbid medical conditions or uncontrolled life threatening infection.
* Patients with recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrythmias are ineligible. Ejection fraction by ECHO must be > 50% and must be performed within 60 days prior to registration, unless the patient has received chemotherapy within that period of time (dexamethasone and thalidomide excluded), in which case the LVEF must be repeated.
* Patients must have a creatinine < 3 mg/dl and a creatinine clearance > 30 ml/minute. Patients with a creatinine clearance of 30-50 ml will only receive a 50% cisplatin dose.
* Patients must have adequate hepatic function defined as serum transaminases < 2 x ULN and direct bilirubin < 2.0 mg/dl.
* Patients must be able to receive full doses of DT PACE, in the opinion of the treating investigator, with the exception of: *Patients that have received prior adriamycin > 450 mg/m2 and LVEF < 55%. Adriamycin will be omitted in these patients; *Patients with a creatinine clearance 30 - 50 ml/minute, who will receive 50% of the cisplatin dose.
* Patients must not have a history of chronic obstructive or chronic restrictive pulmonary disease. Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) > 50% of predicted. Patients unable to complete pulmonary function tests due to myeloma related pain or fracture must have a high resolution CT scan of the chest and must also have acceptable arterial blood gases defined as PO2 greater than 70.

Exclusion Criteria:

* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for at least three years. Prior malignancy is acceptable provided there has been no evidence of disease within the three-year interval.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy test documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2002-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, MD, PhD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Multiple Myeloma — http://www.myeloma.uams.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Waldenstrom's Macroglobulinemia Patients: Participants must have a pathological diagnosis of Waldenstrom's Macroglobulinemia, with advanced and/or symptomatic disease requiring therapy. At least one of the inclusion criteria:
Period: Overall Study
Arm/Group | Waldenstrom's Macroglobulinemia Patients
Started | 12
Completed | 0
Not Completed | 12
Not completed — Physician Decision | 10
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Waldenstrom's Macroglobulinemia Patients
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Response Rates to a Brief Remission Induction Treatment With One or Two Courses of Melphalan-based High-dose Treatment (HDT)
Description: To evaluate the complete and partial response rates, defined in a strict manner, to a brief remission induction treatment with one or two courses of melphalan-based high-dose treatment (HDT) in symptomatic patients with Waldenström's Macroglobulinemia (WM), either untreated or previously treated.
Time Frame: 3 years
Measure: Number; unit: participant
Arm/Group | Waldenstrom's Macroglobulinemia Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Waldenstrom's Macroglobulinemia Patients
Serious Adverse Events (participants affected / at risk) | 6/12
Other Adverse Events (participants affected / at risk) | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Waldenstrom's Macroglobulinemia Patients (N=12)
splenic infarction (General disorders) | 1 (1)
septicemia (Infections and infestations) | 1 (1)
peritonitis (General disorders) | 2 (2)
pneumonia (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Waldenstrom's Macroglobulinemia Patients (N=12)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
dehydration (General disorders) | 1 (1)
nausea, vomiting, diarrhea & fever (Gastrointestinal disorders) | 1 (1)
mucositis (General disorders) | 2 (2)
colitis (Gastrointestinal disorders) | 1 (1)
hypotension (Cardiac disorders) | 1 (1)
septic arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to small numbers of subjects enrolled. Only one participant completed the study. Other participants came off study due to death, toxicity, physician choice, or patient choice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes